CLINICAL TRIAL: NCT00415168
Title: Phase 2 Study of ALIMTA® (Pemetrexed) Plus Cisplatin as First-Line Treatment of Gastric Cancer
Brief Title: Pemetrexed Plus Cisplatin as First-Line Treatment in Stage IV or Recurrence of Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10874; H3E-MW-S108 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed + Cisplatin (Experimental)
  Interventions: Drug: pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: pemetrexed — 700 milligrams/meters squared (mg/m2), intravenous (IV), every 21 days x 6 cycles
  Other Names: LY231514; Alimta
Drug: cisplatin — 75 mg/m2, IV, every 21 days x 6 cycles

SUMMARY:
Study H3E-MW- S108 is a multicenter, single arm, open-label Phase 2 study to determine the response rate of pemetrexed plus cisplatin in patients with Stage IV gastric cancer, not amenable to curative surgery, or recurrence after prior surgery, who have had no prior chemotherapy. It was planned to enroll approximately 50 patients who qualified for tumor response population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the gastric. Stage IV disease, not amenable to curative surgery, or disease recurrence after prior surgery.
* Disease status must be that of measurable disease with presence of at least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* In bidimensionally measurable lesions the longest diameter should be selected for measurement.
* Tumor lesions in areas of prior radiation therapy may be included only if they were clearly progressing.
* If only a single lesion is present in a patient who had prior therapy for gastric adenocarcinoma, the neoplastic nature of the lesion should be confirmed by cytology and/or histology.
* Ultrasound and clinical examination are not allowed for assessment of measurable disease.
* Elevation of tumor markers, pleural or pericardial effusion, ascites, bone lesions, cystic lesions, or carcinomatous lymphangitis pulmonis/cutis is defined as not being measurable.
* Performance Status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Estimated life expectancy of at least 12 weeks.
* No prior chemotherapy or radiotherapy.
* Patient compliance and geographic proximity that allow adequate follow-up.

Adequate organ function including the following:

* Bone marrow: absolute neutrophil count 1.5 x 10 to the ninth power/liter (L), platelets 100 x 10 to the ninth power/L, hemoglobin >=9 grams per deciliter (g/dL).
* Hepatic: bilirubin <=1.5 x upper limit of normal (ULN); alkaline phosphatase, aspartate transaminase and alanine transaminase <=3.0 x ULN.
* Renal: Calculated creatinine clearance >=45 milliliters (ml)/minute.
* Men or women, age 18 to 70 years.
* For women: Must be surgically sterile, post-menopausal, or compliant with a medically approved contraceptive regimen during and for 3 months after the treatment period; must have a negative serum or urine pregnancy test within 7 days before study enrollment and must not be breast-feeding.
* For men: Must be surgically sterile, or compliant with a contraceptive regimen during and for 3 months after the treatment period.
* Signed informed consent from patient.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Concurrent administration of any other tumor therapy.
* Active infection.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Pregnancy.
* Breast-feeding.
* History of significant neurological or mental disorder, including seizures or dementia.
* Have had a prior malignancy other than gastric cancer, carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence.
* Patients with a history of low grade (Gleason score less than or equal to 6) localized prostate cancer will be eligible even if diagnosed less than 5 years previously.
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory drugs 2 days before, the day of, and 2 days after the dose of pemetrexed plus cisplatin.
* If a patient is taking a nonsteroidal anti-inflammatory drug (NSAID) or salicylate with a long half-life it should not be taken 5 days before, the day of, and 2 days after the dose of pemetrexed plus cisplatin.
* Clinically significant ascites or pleural effusion that is apparent at clinical examination and cannot be controlled by drainage or other procedures prior to study enrollment. NOTE: Small effusions noted on computed tomography (CT) scan do not exclude the patient from study enrollment.
* Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.
* Known or suspected brain metastasis. Patients who have clinical signs or symptoms that are suspicious of brain metastasis must have a pretreatment CT or magnetic resonance imaging (MRI) of the brain. A patient with documented brain metastasis, at the time of consideration for study entry or in the past, will be excluded from entering in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) OR 1-317-615-4559 Mon - Fri 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Russia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barnaul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ivanovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol

REFERENCES:
- [Background] United States Food and Drug Administration (US-FDA). 2005. Guidance for Industry: Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics (Draft Guidance). Available at: http://www.fda.gov/cder/guidance/6592dft.htm, accessed 01 November 2005. Currently available at: http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM071590.pdf, accessed 22 June 2010.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 participants signed informed consent and 3 participants were screen failures.
Groups:
- Pemetrexed + Cisplatin: Pemetrexed 700 milligrams/meters squared (mg/m2) plus cisplatin 75 mg/m2, intravenous (IV), every 21 days for 6 cycles
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin
Started | 53
Completed Treatment | 15
Completed | 1
Not Completed | 52
Not completed — Death | 26
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 13
Not completed — Sponsor Decision | 4
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 53
Age Continuous [Mean (Standard Deviation); unit: years] | 54.3 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 53
Region of Enrollment [Number; unit: participants]
  Russian Federation | 53
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — A grading scale is provided for performance status from 0 (fully active, able to carry on all pre-disease performance without restriction) to 5 (dead).
  participants
    0 - Fully Active | 16
    1 - Ambulatory, Restricted Strenuous Activity | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (Objective Response Rate)
Description: Tumor responder is defined as participants exhibiting a best overall study response of complete response (CR; disappearance of all target lesions) or partial response (PR; 30% decrease in sum of longest diameter of target lesions). Non-responders are those who did not meet the above criteria.
Time Frame: Baseline to time of response up to six or eight 21-day cycles of treatment
Population: All patients enrolled in the study with a histologically confirmed diagnosis of adenocarcinoma of the gastric, disease status of measurable disease with presence of at least 1 measurable lesion, with no concurrent administration of any other tumor therapy or known or suspected brain metastasis who received at least 1 dose of study therapy.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 53
percentage of responders
  Responder | 32.1 [19.9 to 46.3]
  Non-Responder | 67.9 [53.7 to 80.1]

2. Secondary Outcome: Duration of Response
Description: Measured from the time of first documentation of CR or PR (whichever status is first recorded) until the date of time to disease progression.
Time Frame: Time of response to progressive disease up to six or eight 21-day cycles of treatment; maximum duration of study follow-up was 17.4 months
Population: Full Analysis Set: This analysis set includes all data from all patients receiving at least one dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 53
months | 3.8 [3.3 to 4.7]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as time from baseline to the date of disease progression or death on study, whichever occurs first. The PFS 1 definition from the United States Food and Drug Administration (FDA) draft guidance on clinical endpoints was used (FDA 2005).
Time Frame: Baseline to measured progressive disease or death up to six or eight 21-day cycles of treatment; maximum duration of study follow-up was 17.4 months
Population: Full Analysis Set: This analysis set includes all data from all patients receiving at least one dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 53
months | 3.7 [2.7 to 5.2]

4. Secondary Outcome: Overall Survival
Description: Defined as the time from baseline to date of death due to any cause. Survival time is censored at the date of last contact for patients who are still alive or lost to follow up.
Time Frame: Baseline to date of death from any cause up to six or eight 21-day cycles of treatment; maximum duration of study follow-up was 17.4 months
Population: Full Analysis Set: This analysis set includes all data from all patients receiving at least one dose of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 53
months | 8.8 [6.0 to 9.5]

5. Secondary Outcome: Number of Participants With Pharmacology Toxicity - Grade 3 or 4 Laboratory Toxicity Possibly Related to Study Therapy
Description: Common toxicity criteria (CTC) Grade 3 (severe) or 4 (life-threatening or disabling) laboratory toxicity possibly related to study therapy. A grading (severity) scale is provided for each event term. Grades range from 0 (none) to 5 (death).
Time Frame: Baseline through six or eight 21-day cycles of treatment, up to 30 days after study drug discontinuation
Population: Full Analysis Set: This analysis set includes all data from all patients receiving at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 53
participants
  Any Grade 3 or 4 Laboratory Toxicity | 29
  Bone/Blood Marrow - Other | 1
  Lymphopenia | 1
  Platelets | 4
  Hemoglobin | 6
  Leukocytes (Total White Blood Cells) | 15
  Neutrophils/Granulocytes | 29
  Uric Acid Serum-High | 1
  Metabolic/Laboratory - Other | 3

6. Secondary Outcome: Number of Participants With Pharmacology Toxicity - Grade 3 or 4 Non-Laboratory Toxicity Possibly Related to Study Therapy
Description: Common toxicity criteria (CTC) Grade 3 (severe) or 4 (life-threatening or disabling) non-laboratory toxicity possibly related to study therapy. A grading (severity) scale is provided for each event term. Grades range from 0 (none) to 5 (death).
Time Frame: Baseline through six or eight 21-day cycles of treatment, up to 30 days after study drug discontinuation
Population: Full Analysis Set: This analysis set includes all data from all patients receiving at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 53
participants
  Any Grade 3 or 4 Non-Laboratory Toxicity | 5
  Anorexia | 1
  Diarrhea | 1
  Renal Failure | 1
  Vomiting | 1
  Nausea | 2
  Fatigue | 3

7. Secondary Outcome: Number of Participants Who Died During the Study
Time Frame: During study drug therapy up to six or eight 21-day cycles or treatment; maximum duration of study follow-up was 17.4 months
Population: Full Analysis Set: This analysis set includes all data from all patients receiving at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 53
participants
  Study Disease | 18
  Cardiac Failure Acute | 1
  Death (General Disorders/Administration Site Cond) | 1
  Intestinal Hemorrhage | 1
  Pancytopenia | 1
  Sudden Death | 3
  Multi-Organ Failure | 1

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 9/53
Other Adverse Events (participants affected / at risk) | 49/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=53)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Sudden death (General disorders) | 3 (3)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=53)
Anaemia (Blood and lymphatic system disorders) | 10 (10)
Leukopenia (Blood and lymphatic system disorders) | 13 (34)
Neutropenia (Blood and lymphatic system disorders) | 30 (67)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 14 (45)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 9 (12)
Fatigue (General disorders) | 13 (26)
Pyrexia (General disorders) | 5 (5)
Creatinine renal clearance decreased (Investigations) | 3 (4)
Haemoglobin decreased (Investigations) | 10 (13)
Neutrophil count decreased (Investigations) | 8 (14)
Platelet count decreased (Investigations) | 8 (9)
Weight decreased (Investigations) | 5 (5)
White blood cell count decreased (Investigations) | 11 (18)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days